CLINICAL TRIAL: NCT00005749
Title: Project Andale--Increasing Exercise in Hispanic Women
Status: Completed | Type: Observational
Sponsor: San Diego State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5061; R18HL052704 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To determine the differential effectiveness of a culturally tailored program to shape and maintain moderate intensity physical activity and to improve cardiorespiratory fitness among low SES sedentary Latino women.

DETAILED DESCRIPTION:
BACKGROUND:

Latino women are at high risk for cardiovascular (CVD) and other chronic diseases, in part, due to sedentary lifestyle, obesity, and poor fitness. Few studies assess long-term physical activity, fewer observe maintenance and none have demonstrated effective procedures for sustaining exercise. Only one study has demonstrated increased moderate exercise and none has demonstrated maintenance of physical activity among Latino women. Theoretically-based procedures (shaping, contingency management, relapse prevention, and social reinforcement) hypothesized as necessary to maintain physical activity had not yet been tested experimentally.

DESIGN NARRATIVE:

The 210 Latinas were assigned at random to one of three groups: one six month physical activity intervention, one physical activity plus maintenance intervention, and one safety education control. Exercise training emphasized walking. Bilingual exercise leaders, aided by peer models from the community, used shaping procedures to establish daily walking in participants. In the maintenance program, family incentives reinforced transfer to community exercise and were used to establish positive feedback loops to promote activity within the family. Peer led community exercise sessions, and community activism were also used to establish social networks which reinforced sustained physical activity.

Program support was faded out as naturally occurring social support for Community exercise was established. Four (baseline, post-intervention, post-maintenance, follow-up), repeated measures over 24 months assessed fitness (VO2max), physical activity (PAR), and CVD risk factors. Theoretically important mediating variables, such as self-efficacy, social support, stage of change for exercise, decisional balance, and home exercise environment were explored. Repeated measures analyses were used to determine significant differences among groups, time and group by time main effects. This study was the first to attempt to engineer maintenance of physical activity among minority women. Results will provide a model to be used to sustain physical activity and reduce the risk of cardiovascular and other diseases. If effective, this analysis will also serve as a model for designing programs to sustain physical activity in the increasingly sedentary general population.

The study was renewed in January 2000 to continue through December 2001.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-07; Study Completion 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Melbourne Hovell — San Diego State University